CLINICAL TRIAL: NCT02487173
Title: A Prospective Multi-Centre Study of the Respirio Flu Test Performance Versus Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) and Sofia® Influenza A+B Fluorescent Immunoassay (FIA) for the Rapid Detection of Influenza A/B
Brief Title: Validation of the Respirio Flu Test for the Rapid Identification of Influenza A/B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellume Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RESP15001
Record Dates: First submitted 2015-06-26; First posted 2015-07-01 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Influenza A; Influenza B
MeSH Terms: interventions — Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respirio Flu Test (Experimental): Upper respiratory tract samples from participants will be tested with:
  * Respirio Flu Test
  * Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)
  * Sofia® Influenza A+B Fluorescent Immunoassay (FIA)
  Interventions: Device: Respirio Flu Test; Device: Reverse Transcriptase Polymerase Chain Reaction (RT-PCR); Device: Sofia® Influenza A+B Fluorescent Immunoassay (FIA)

INTERVENTIONS:
Device: Respirio Flu Test — The Respirio Flu Test is a rapid test for the detection of influenza A or influenza B in nasal secretions. The Respirio Flu Test is designed to be simple to use and generates a result within 20 minutes.
Device: Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) — Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) is a molecular diagnostic technique for the detection and identification of influenza viruses, both for clinical samples and isolates. The reverse-transcriptase polymerase chain reaction (RT-PCR) allows template viral RNA to be reverse transcribed producing complementary DNA (cDNA) which can then be amplified and detected.
Device: Sofia® Influenza A+B Fluorescent Immunoassay (FIA) — Sofia® Influenza A+B Fluorescent Immunoassay (FIA) employs immunofluorescence to detect influenza A and influenza B viral nucleoprotein antigens in nasal swab, nasopharyngeal swab, and nasopharyngeal aspirate/wash samples taken directly from symptomatic patients.

SUMMARY:
The primary purpose of this study is to validate the sensitivity and specificity of the Respirio Flu Test in detecting Influenza A, when used by subjects, as compared to the gold standard for detection, Reverse Transcriptase Polymerase Chain Reaction (RT-PCR).

The secondary aims are to:

* validate the sensitivity and specificity of the Respirio Flu Test in detecting Influenza B , when used by subjects, as compared to the gold standard for detection, Reverse Transcriptase Polymerase Chain Reaction (RT-PCR).
* assess agreement (positive and negative) between Respirio Flu Test and Sofia® Influenza A+B Test in detecting Influenza A;
* assess agreement (positive and negative) between Respirio Flu Test and Sofia® Influenza A+B Test in detecting Influenza B;
* evaluate the correct interpretation of the Respirio Flu Test results by subjects with Influenza-like illness symptoms;
* evaluate the subjects' satisfaction with the convenience, comfort and ease of use of the Respirio Flu Test;
* evaluate the subjects' comprehension of the Respirio Flu Test labelling; and
* establish the minimum sample weight required to achieve a result with the Respirio Flu Test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 1 year;
* Rhinorrhea;
* ≤ 72 hours from onset of Influenza-like illness symptoms;
* Subject (or parent/legal guardian) capable and willing to give informed consent/assent.
* Subject (or parent/legal guardian) able to read and write in English.

Exclusion Criteria:

* Has undergone treatment with antivirals within the previous 7 days;
* Has been vaccinated by means of an Influenza nasal spray/mist vaccine within the previous 7 days;
* Recent craniofacial injury or surgery, including surgery to correct deviation of the nasal septum, within the previous 6 months;
* Currently enrolled in another clinical trial or used any investigational device within 90 days preceding informed consent;
* Has had prior exposure to the Respirio Flu Test;
* Subject (or parent/legal guardian) residing at the same residential address as a subject currently enrolled in this study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Of participants positive for influenza A by ReverseTranscriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza A by Respirio Flu Test. | Day 1
  Establish sensitivity against a gold standard. Report as a percentage of participants with 95% confidence limits.
Of participants negative for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza A by Respirio Flu Test. | Day 1
  Establish specificity against a gold standard. Report as a percentage of participants with 95% confidence limits.

SECONDARY OUTCOMES:
Of participants positive for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza B by Respirio Flu Test. | Day 1
  Establish sensitivity against a gold standard. Report as a percentage of participants with 95% confidence limits.
Of participants negative for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza B by Respirio Flu Test. | Day 1
  Establish specificity against a gold standard. Report as a percentage of participants with 95% confidence limits.
Percent of participants positive for influenza A by Sofia® Influenza A+B Test and Respirio Flu Test. | Day 1
  Establish positive agreement against an imperfect standard. Report as a percentage of participants with 95% confidence limits.
Percent of participants negative for influenza B by Sofia® Influenza A+B Test and Respirio Flu Test. | Day 1
  Establish negative agreement against an imperfect standard. Report as a percentage of participants with 95% confidence limits.
Combine positive and negative agreement of Respirio Flu Test and Sofia® Influenza A+B Test to establish overall agreement. Report as a percentage of participants with 95% confidence limits. | Day 1
Percent of participants who correctly interpret result of Respirio Flu Test. | Day 1
  Agreement between trained staff and participants. Report as a percentage of participants with 95% confidence limits.
Scores from questionnaire to assess ease of use, comfort and convenience of Respirio Flu Test. | Day 1
  The ease of use questionnaire will provide the following:
  • Total number of responses to each question and the percentage of participants selecting each response (most on a 5 point Likert scale).
Percent of participants correctly determining eligibility and conditions for use of Respirio Flu Test from scores on a label comprehension questionnaire. | Day 1
  The label comprehension questionnaire will provide the following data
  * Total number of responses to the question and the percentage of participants selecting each option.
  * Number and percentage of participants selecting the correct answer to each question.
  * Overall percentage of patients with an acceptable level of comprehension.
Weight of sample deposited in Respirio Flu Test. | Day 1
  Establish minimum weight of sample required to obtain a valid result from the Respirio Flu Test.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Taringa 7 Day Medical Practice, Brisbane, Queensland
  - Graceville Medical, Brisbane, Queensland
  - Inala Primary Care, Brisbane, Queensland
  - Limestone Medical Centre, Ipswich, Queensland